CLINICAL TRIAL: NCT04912661
Title: Iron and Vaccine-preventable Viral Disease - an Experimental Study
Brief Title: Iron and Vaccine Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Principal Investigator, Nicole Stoffel, PhD, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DIVA I
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Iron Deficiency Anemia; Vaccine Preventable Disease; Vaccine Response Impaired; Iron Deficiency Anemia Treatment
MeSH Terms: conditions — Anemia, Iron-Deficiency; Vaccine-Preventable Diseases | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate iron treatment (Active Comparator): intravenous iron carboxymaltose before vaccination
  Interventions: Dietary Supplement: Ferinject
- No iron treatment (No Intervention): no intravenous iron carboxymaltose before vaccination

INTERVENTIONS:
Dietary Supplement: Ferinject — intravenous iron carboxymaltose
  Arms: Immediate iron treatment

SUMMARY:
Vaccines often underperform in Africa compared to high-income countries. Why vaccines do not work as well in Africa remains uncertain. Malnutrition likely plays a role. Our study objective is to assess whether iron deficiency anaemia in young women impairs their immune response to viral vaccines, and whether iron treatment improves their response.

DETAILED DESCRIPTION:
Group 1 (immediate iron treatment) will receive iron treatment before vaccination. Women in both groups will receive two intramuscular vaccines (influenza and yellow fever). Vaccine response will be measured 28 and 56 days after vaccine administration in both groups. Group 2 (delayed iron treatment) will receive iron treatment at study end.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Zinc protoporphyrin > or equal 40 mmol/mol heme
* hemoglobin < or equal 109 g/L
* no malaria
* no known HIV infection
* no medical condition that precludes study involvement
* no iron supplementation 1 week prior to study start
* no recent tuberculosis infection
* no vaccination of yellow fever or influenza prior to enrolment
* not pregnant

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Antibody titers | at 35 days
Antibody titers | at 63 days
Seroconversion | at 35 days
Seroconversion | at 63 days
Antibody avidity Index | at 35 days
  percentage of antibodies that remain bound to beads
Antibody avidity Index | at 63 days
  percentage of antibodies that remain bound to beads

SECONDARY OUTCOMES:
antiviral immunoglobulin G response | day 0
  Immunoassay
antiviral immunoglobulin G response | day 7
  Immunoassay
antiviral immunoglobulin G response | day 35
  Immunoassay
antiviral immunoglobulin G response | day 63
  Immunoassay
immune cell populations | day 0
  number and type of immune cells
immune cell populations | day 7
  number and type of immune cells
immune cell populations | day 35
  number and type of immune cells
immune cell populations | day 63
  number and type of immune cells
Proteomics | day 0
  Proteins involved in immune response
Proteomics | day 7
  Proteins involved in immune response
Proteomics | day 35
  Proteins involved in immune response
Proteomics | day 63
  Proteins involved in immune response
Transcriptomics | day 0
  Genes involved in immune response
Transcriptomics | day 7
  Genes involved in immune response
Transcriptomics | day 35
  Genes involved in immune response
Transcriptomics | day 63
  Genes involved in immune response
Immune cell cytokine secretion | day 7
  ELISpot
Immune cell cytokine secretion | day 35
  ELISpot
Hemoglobin | day 0
  iron status parameter
Hemoglobin | day 7
  iron status parameter
Hemoglobin | day 35
  iron status parameter
Hemoglobin | day 63
  iron status parameter
Plasma Ferritin | day 0
  iron status parameter
Plasma Ferritin | day 7
  iron status parameter
Plasma Ferritin | day 35
  iron status parameter
Plasma Ferritin | day 63
  iron status parameter
Transferrin receptor | day 0
  iron status parameter
Transferrin receptor | day 7
  iron status parameter
Transferrin receptor | day 35
  iron status parameter
Transferrin receptor | day 63
  iron status parameter
Transferrin saturation | day 0
  iron status parameter
Transferrin saturation | day 7
  iron status parameter
Transferrin saturation | day 35
  iron status parameter
Transferrin saturation | day 63
  iron status parameter
C-reactive protein | day 0
  inflammation status parameter
C-reactive protein | day 7
  inflammation status parameter
C-reactive protein | day 35
  inflammation status parameter
C-reactive protein | day 63
  inflammation status parameter
Alpha-glycoprotein | day 0
  inflammation status parameter
Alpha-glycoprotein | day 7
  inflammation status parameter
Alpha-glycoprotein | day 28
  inflammation status parameter
Alpha-glycoprotein | day 56
  inflammation status parameter
retinol binding protein | day 0
  marker for Vitamin A status
retinol binding protein | day 7
  marker for Vitamin A status
retinol binding protein | day 35
  marker for Vitamin A status
retinol binding protein | day 63
  marker for Vitamin A status
plasma zinc | day 0
plasma zinc | day 7
plasma zinc | day 35
plasma zinc | day 63

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stoffel, PhD, Principal Investigator — ETH Zurich
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: No